CLINICAL TRIAL: NCT06533605
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, and Initial Efficacy of SSGJ-706 Monotherapy for Patients With Advanced Solid Tumors
Brief Title: Phase I Clinical Study to Evaluate the Safety and Efficacy of SSGJ-706 Monotherapy for Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-706-101
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors Patients
Keywords: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Arm 1 (Experimental): dose level 1 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 2 (Experimental): dose level 2 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 3 (Experimental): dose level 3 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 4 (Experimental): dose level 4 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 5 (Experimental): dose level 5 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 6 (Experimental): dose level 6 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 7 (Experimental): dose level 1 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 8 (Experimental): dose level 2 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 9 (Experimental): dose level 3 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 10 (Experimental): dose level 4 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 11 (Experimental): dose level 5 of SSGJ-706
  Interventions: Drug: SSGJ-706
- Arm 12 (Experimental): dose level 6 of SSGJ-706
  Interventions: Drug: SSGJ-706

INTERVENTIONS:
Drug: SSGJ-706 — Bispecific antibody

SUMMARY:
This study includes two parts, different part has different administration frequencies of SSGJ-706.

DETAILED DESCRIPTION:
This study is a study of SSGJ-706 monotherapy in advanced Solid Tumors. This study includes two parts, different part has different administration frequencies of SSGJ-706. Part A is QW and part B is Q3W. Each part will assess the efficacy and safety of the preset several dose levels of SSGJ-706 in advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented advanced or metastatic Solid Tumors .
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >=3 months.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to SSGJ-706 The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
DLTs | 12 months
  Dose limiting toxicity
MTD or MAD | 12 months
  maximum tolerated dose or the maximum administered dose if MTD is not reached

SECONDARY OUTCOMES:
The blood concentration of SSGJ-706 | 12 months
  PK characteristics

IPD SHARING:
Plan to Share IPD: No